CLINICAL TRIAL: NCT06053671
Title: Dissecting mTOR Pathway Mosaicism in FCDII-Harbouring Epileptic Brain and Peripheral Tissue.
Brief Title: Mos-FED (Mosaicism in Focal Epilepsy Cortical Dysplasia Tissue)
Acronym: MosFED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Danish Epilepsy Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 303113_28022022; 22/WA/0326 (Other: Research Ethics Committee (UK))
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Focal Cortical Dysplasia; Epilepsy
MeSH Terms: conditions — Focal Cortical Dysplasia; Epilepsy | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with histologically confirmed FCDIIA/B undergoing or post Epilepsy Surgery (Experimental): Genetic screening of DNA samples (blood, mucosal swab, brain tissue)
  Interventions: Genetic: Blood and nasal swab sampling

INTERVENTIONS:
Genetic: Blood and nasal swab sampling — Genetic screening of DNA samples (blood, mucosal swab, brain tissue) from 60-100 patients with histologically confirmed diagnosis of FCDIIA/B identified from Epilepsy Surgery Databases.
  Other Names: Analysis of Epilepsy Surgical tissue

SUMMARY:
Focal cortical dysplasia (FCD) is a malformation of brain development, the most common cause of drug-resistant epilepsy and often caused by mutations in mammalian target of rapamycin (mTOR) pathway genes. Patients with FCD develop drug-resistant seizures. This study will look at FCD tissue removed during epilepsy surgery and aims to detect mutations in mTOR pathway genes in brain cells. Secondly, the investigators will establish if evidence of mutations found in brain cells can also be detected as circulating free DNA (cfDNA) in blood. By looking at which genes are made into proteins in individual cells found in epilepsy surgical tissue (single cell expression profiling),the investigators will attempt to identify new genetic targets in FCD.

The main outcome will be finding new causes of epilepsy with FCD and the development of new diagnostic and screening tools.

DETAILED DESCRIPTION:
Primary Objectives:

1. To identify if somatic mosaicism for mTOR is present in resected tissue from patients with FCDIIA/B, and can be detected in DNA from patient's serum as circulating free DNA (cfDNA) or from nasal epithelial cells collected non-invasively by olfactory mucosal brush swab.
2. To establish if single cell expression profiling from resected fresh frozen tissue reveals novel FCD causing pathways and single cell RNA sequencing increases the yield of mTOR pathway variant detection.
3. To determine if phosphorylated upstream and downstream mTOR pathway components can be characterised by immunohistochemistry and Western blot as novel biomarkers of mTOR activation in human FCDII tissue.

Secondary Objectives:

To engage with patients, representatives and charitable organisations to assess feasibility and develop plan to set up a future trial of mTOR inhibitor treatment.

ELIGIBILITY:
Epilepsy in Focal Cortical Dysplasia Type IIA/B

Key Inclusion Criteria:

1. Adult and Paediatric Patients (male and female)
2. A histologically proven diagnosis of FCDIIA/B or a suspected diagnosis of FCDIIA/B (on MRI/EEG and PET grounds) awaiting resective Epilepsy surgery.
3. Able to attend appointment/hospital and undergo sampling of serum and nasal swab
4. Informed Consent Available

   Key Exclusion Criteria:
5. Any acute or chronic conditions that could limit the ability of the patient to participate in the study.
6. Refusal to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-09 (Actual); Primary Completion 2025-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
somatic mosaicism | 2 years
  This study will measure and report the rate of somatic mosaicism for mTOR pathway genes in resected brain tissue and peripheral blood and nasal mucosal cells from patients with FCDIIA/B assessed by panel genetic sequencing of genomic and free circulating DNA .
single cell expression profiling | 2 years
  This study will measure and report novel FCD causing mutations through single cell expression profiling from resected fresh frozen tissue.
phosphorylated targets | 2 years
  This study will measure phosphorylation of upstream and downstream mTOR pathway components by immunohistochemistry and Western blot in human FCDII tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised clinical data associated with the tissue will be deposited with the King's Open Research Data System (KORDS), a trusted research environment, which meets UKRI data retention and sharing requirements. KORDS also enables published datasets to be long-term discoverable, accessible and citable
Supporting Information: CSR
Time Frame: Data will be accessible to others outside of our team once published or within three years of the end of the grant, to allow for completion of publications and project proposals.
Access Criteria: Governance Digital data available to the wider community will be controlled by KORDS application procedures. Before any data are published, we will conduct a Data Protection Impact Assessment (DPIA) in accordance with the UK GDPR. Requests for unpublished and/or genomic data will be controlled by a Data Management Committee. Data and Biological Material Transfer and Sharing Agreements which defines the scope of use, timeline and further distribution limits will be agreed.
  Data will be accessible to others outside of our team once published or within three years of the end of the grant, to allow for completion of publications and project proposals.
  We will attempt to limit restriction to human data sharing by gaining participant's consent for data sharing, and by anonymising data. Our consent form will clearly describe proposed data sharing schemes, their benefits and potential risks, whilst safeguarding participants.